

### Protocol for observational studies based on existing data

| Document Number: | c03412460-01 |
|---|---|
| BI Study Number: | 1160-0235 |
| BI Investigational Product(s): | Dabigatran etexilate (Pradaxa®) |
| Title: | Pradaxa Initiation Post-Stroke Study: SITS-Pradaxa 1. A retrospective analysis from the SITS-AF Registry on treatment initiation of dabigatran etexilate in non-valvular atrial fibrillation patients hospitalized with acute ischemic stroke |
| Lay Title | This study uses the SITS Registry to find out when patients with a heart rhythm disorder (atrial fibrillation) start treatment with dabigatran after they had a stroke |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | 05 July 2017 |
| PASS: | No |
| EU PAS register number: | EUPAS17165 |
| Active substance: | B01AE07 - dabigatran etexilate (Pradaxa® ) |
| Medicinal product: | Dabigatran etexilate |
| Product reference: | EU/1/08/442/001-019 |
| Procedure number: | EMEA/H/C/000829 |
| Joint PASS: | No |
| Research question and objectives: | <ul> <li>Primary Objective:</li> <li>To evaluate the timing of dabigatran treatment initiation in patients with non-valvular atrial fibrillation (NVAF) after hospitalization for first ever ischaemic stroke (the index event) in order to prevent secondary stroke.</li> <li>Secondary Objectives:</li> <li>To describe baseline characteristics for patients</li> </ul> |

c03412460-01

| | treated with dabigatran according to time of dabigatran initiation. |
|---|---|
| | <ul> <li>To describe self-reported factors important for the<br/>physician's decision as to the time of dabigatran<br/>initiation in the post-ischemic stroke setting.</li> </ul> |
| | <ul> <li>To describe self-reported factors important for<br/>physician's decision as to which dabigatran dose was<br/>used in the post-ischemic stroke setting.</li> </ul> |
| <b>Countries of study:</b> | Data from all patients in European countries* actively registered in the SITS Registry until 31 July 2018, will be considered for analysis. |
| | (*countries such as, Italy, United Kingdom, Czech<br>Republic, Sweden, Germany, Poland, Spain, Finland,<br>Portugal, Slovakia, Denmark, Estonia, Norway Belgium,<br>Hungary, Slovenia, Croatia, Austria, Lithuania, France,<br>Greece, Netherlands, Ireland, Ukraine and Iceland) |
| Authors: | |
| | E-mail: |
| | E-mail: |
| | Address: |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | _ |
|---|---|
| | Phone: Fax: |
| | Trial Clinical Monitor |
| | Phone Fax |
| | E-mail: |
| Marketing authorisation holder: | |
| MAH contact person: | |
| Date: | 05 July 2017 |
| | Page 1 of 42 |
| Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. | |
| This document may not | t - in full or in part - be passed on, reproduced, published or |

otherwise used without prior written permission

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 1. TABLE OF CONTENTS

| TITI | E PAGE |
|------|---------------------------------------------|
| 1. | TABLE OF CONTENTS |
| | LIST OF ABBREVIATIONS |
| | RESPONSIBLE PARTIES |
| 4. | ABSTRACT |
| 5. | AMENDMENTS AND UPDATES |
| 6. | MILESTONES |
| 7. | RATIONALE AND BACKGROUND |
| 8. | RESEARCH QUESTION AND OBJECTIVES |
| 9. | RESEARCH METHODS |
| 9.1 | STUDY DESIGN |
| 9.2 | SETTING |
| 9.3 | VARIABLES |
| 9. | 3.1 Exposures |
| 9 | .3.2 Outcomes |
| | 9.3.2.1 Primary outcomes |
| | 9.3.2.2 Secondary outcomes |
| | 19 |
| 9 | .3.3 Covariates |
| 9.4 | DATA SOURCES |
| 9.5 | STUDY SIZE21 |
| 9.6 | DATA MANAGEMENT |
| 9.7 | DATA ANALYSIS |
| 9. | .7.1 Main analysis |
| | 23 |
| | .7.3 Interim analysis |
| 9.8 | QUALITY CONTROL 24 |
| 9.9 | LIMITATIONS OF THE RESEARCH METHODS |
| 9.10 | - |
| 9.11 | .10.1 Ethical approval and informed consent |
| | PIAS 26 |

c03412460-01

| 10. | PROTECTION OF HUMAN SUBJECTS | 27 |
|---|---|---|
| 11. | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 28 |
| 12. | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY | |
| | RESULTS | 29 |
| 13. | REFERENCES | 30 |
| 13. | 1 PUBLISHED REFERENCES | 30 |
| 14. | APPENDICES | 33 |
| Apj | pendix 1: CHADS <sub>2</sub> Stroke Risk Score | 33 |
| App | pendix 2: CHA <sub>2</sub> DS <sub>2</sub> -VAS <sub>c</sub> Stroke Risk Score | 34 |
| Apj | pendix 3: HAS-BLED Bleeding Risk SCORE | 35 |
| App | pendix 4: List of stand-alone documents | 36 |
| App | pendix 5: ENCePP checklist for study protocols | 37 |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 2. LIST OF ABBREVIATIONS

AE Adverse Event AF Atrial Fibrillation

CHAD<sub>2</sub> score Stroke Risk score based on a point system, which includes history of

Congestive heart failure, Hypertension, Age (≥ 75), Diabetes

mellitus, Stroke/TIA.

CHA<sub>2</sub>DS<sub>2</sub>- Stroke Risk score based on a point system, which includes history of

VASc score Congestive heart failure, Hypertension, Age ( $\geq 75$ ), Diabetes

mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex category

CI Confidence Interval

EMA European Medicines Agency

ENCePP European Network of Centers for Pharmacoepidemiology and

Pharmacovigilance

EUPAS The European Union electronic Register of Post-Authorisation

Studies (EU PAS Register)

GVP Good Pharmacovigilance Practices

HAS-BLED Bleeding Risk score based on a point system, which includes

Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years),

Drugs and Alcohol

ICO International Coordinating Office (at SITS International)

IEC Independent Ethics Committee
INR International Normalized Ratio
IRB Institutional Review Board

LV EF Left Ventricular Ejection Fraction MAH Marketing authorisation holder

MI Myocardial Infarction mRS modified Rankin Scale

N.A. Not applicable

NIHSS National Institute of Health Stroke Scale NOAC Non-vitamin K Oral Anticoagulation NVAF Non-valvular Atrial Fibrillation

OAC Oral Anticoagulant

p.o. per os (oral)

PASS Post-Authorisation Safety Study

q.d. quaque die (once a day)

SITS Safe Implementation of Treatment in Stroke (Registry)

SITS-MOST Safe Implementation of Thrombolysis in Stroke-Monitoring Study

SmPC Summary of Product Characteristics

TCM Trial Clinical Monitor
TIA Transient Ischaemic Attack
t.i.d. ter in die (3 times a day)

TMF Trial Master File

TMM Team Member Medicine VKA Vitamin K Antagonist

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. RESPONSIBLE PARTIES

### **SITS International**

Study coordinator:

Study advisor:

Study administrative operator:

SITS Executive Assistant:

Database

SITS User Service and IT

Network and Research Executive:

### **Boehringer Ingelheim**

Team Member Medicine (TMM):

Trial Clinical Monitor (TCM):

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4. ABSTRACT

| | | T | 1 |
|---|---|---|---|
| Name of company | : | | |
| Boehringer Ingelheim | | | |
| Name of finished a<br>product:<br>Pradaxa | nedicinal | | |
| Name of active ing<br>Dabigatran etexilate | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 05 July 2017 | 1160-0235 | 1.0 | N.A. |
| Title of study: | retrospective a<br>Registry on tre | ion Post-Stroke Study: SITS-<br>nalysis of existing data from<br>eatment initiation of dabigatra<br>fibrillation patients hospitaliz<br>e | the SITS-AF<br>an etexilate in non- |
| Rationale and background: | Dabigatran etexilate (Pradaxa) is the first non-VKA oral anticoagulant (NOAC) for stroke prevention in non-valvular atrial fibrillation (NVAF) patients. Compared with warfarin, dabigatran 150 mg twice daily exhibited lower rates of stroke and systemic embolism, but similar rates of major haemorrhage; whereas treatment with dabigatran 110 mg twice daily showed similar rates of stroke and systemic embolism, but lower rates of major haemorrhage. Both dosages of dabigatran etexilate were associated with lower rates of intracranial haemorrhage. | | |
| | including Euro<br>systemic embo<br>results from the<br>of anticoagular<br>been confirmed<br>severe, disabling<br>stroke within the | s been approved in most count<br>ope and US to reduce the risk<br>olism in patients with NVAF.<br>e RE-LY study concerning that<br>therapy with dabigatran in<br>d in routine clinical practice of<br>any stroke within the previous<br>the previous 14 days was exclude<br>te setting on secondary stroke | of stroke and In addition, the ne use and outcome NVAF patients have data. In RE-LY, 6 months, or any luded and therefore, |
| | ischemic stroke its use and is b | of warfarin for the secondary<br>e in NVAF has been establish<br>ased on the severity of the in<br>ays for TIA up to 3-4 weeks f | hed over the years of dex event. It ranges |

c03412460-01

| Name of company | 7.• | | |
|---|---|---|---|
| Name of finished medicinal product: Pradaxa | | | |
| Name of active ing<br>Dabigatran etexilat | _ | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 05 July 2017 | 1160-0235 | 1.0 | N.A. |
| | | bigatran the time ranges of in ve not yet been established. | itiation after the |
| | dabigatran etex | aim of this study is to explor<br>xilate for stroke prevention in<br>setting in routine clinical pra | NVAF patients in |
| | approximately | he SITS Registry the entered 1000 eligible patients, that in event, will be extracted for r | nitiated dabigatran |
| Research question and objectives: | <ul> <li>Primary Objective:</li> <li>To evaluate the timing of dabigatran treatment initiation in patients with non-valvular atrial fibrillation (NVAF) the after hospitalization for first ever ischaemic stroke, in order to prevent secondary stroke.</li> </ul> | | |
| | Secondary Ob | ojectives: | |
| | <ul> <li>dabigatran</li> <li>To describe physician's the post-iso</li> <li>To describe decision as</li> </ul> | e baseline characteristics for according to time of dabigate e self- reported factors imports decision as to the time of datachemic stroke setting. The self- reported factors imports to which dabigatran dose was troke setting. | ran initiation. tant for the abigatran initiation in tant for physician's |

c03412460-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelh | neim | | |
| Name of finished medicinal product: Pradaxa | | | |
| Name of active ing<br>Dabigatran etexilat | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 05 July 2017 | 1160-0235 | 1.0 | N.A. |
| Study design: | This is a retros from the SITS | pective observational study registry | using existing data |
| Population: | NVAF patients stroke. | s presenting with their first ev | er ischemic acute |
| Variables: | <ul> <li>Patient characteristics such as age, stroke severity based on NIHSS, selected comorbidities, CHADS<sub>2</sub>, CHA<sub>2</sub>DS<sub>2</sub>-VAS<sub>c</sub> and bleeding (HAS-BLED) risk scores, prior oral anticoagulation treatment (dabigatran, Factor Xa Inhibitors, VKA) at index stroke date, the timing of dabigatran treatment initiation for secondary prevention of stroke when initiated within 3 months.</li> <li>Physicians' self-reported factors important for their decisions when to initiate dabigatran in the post-ischemic stroke setting and factors important for physician's decision which dabigatran dose is used in the post-ischemic stroke setting for prevention of stroke in NVAF.</li> </ul> | | |
| Data sources: | treated patients | stry data of approximately 10 s in European countries registrated by 31 st July 2018). | _ |
| Study size: | | v 1000 NVAF patients who as xilate within 3 months of their | |

c03412460-01

| | | T | |
|---|---|---|---|
| Name of company: | | | |
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Pradaxa | | | |
| Name of active ing<br>Dabigatran etexilate | • | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 05 July 2017 | 1160-0235 | 1.0 | N.A. |
| | , | event) constitute the main and | |
| Data analysis: | Descriptive statistics (absolute numbers and relative frequencies, means, standard deviations, medians, inter quartile ranges, minimum and maximum values, 95% confidence intervals and proportions, as appropriate) for baseline and demographic characteristics for all included patients will be provided as appropriate for the variable of interest. | | |
| | • | ysis will focus on NVAF pati<br>acute stroke and treated with<br>ex event. | 1 0 |
| | for secondary p | be the timing of dabigatran to<br>prevention of stroke when treats in the post-stroke setting. | |
| | the Registry us<br>physician's dec<br>and the self-reg<br>dose is used in<br>of stroke. Desc | arize the self- reported factor<br>sing a dedicated question) im-<br>cision for the timing when to<br>ported factors important for we<br>the post-ischemic stroke setteriptions will also be stratified<br>nitiation if sample size allow | portant for the initiate dabigatran which dabigatran ing for prevention d according to time |
| | dabigatran trea<br>prevalent NVA | ients will be described stratifutment initiation, newly diagnaF, prior treatment with anticulation therapy, stroke seve | osed NVAF or oagulation including |

c03412460-01

| Name of company | • | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Pradaxa | | | |
| Name of active ing<br>Dabigatran etexilate | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 05 July 2017 | 1160-0235 | 1.0 | N.A. |
| | | dose of dabigatran, if the sam | |
| | | ent safety related informationg this study. Thus, individual | |
| Milestones: | since the prese<br>fibrillation and<br>After approxin<br>European Cent | ent data are collected in the Sentation of 'Extended data ental oral anticoagulant', 1 <sup>st</sup> July in ately 1000 dabigatran treated tres are registered in SITS-Alla will be extracted and a retroe performed. | ry option for atrial 2014. d patients from F (expected by July |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. AMENDMENTS AND UPDATES

Not applicable

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. MILESTONES

| Milestone | Planned Date |
|---|---|
| Start of study/data collection | 17 July 2017 |
| End of data collection | 31 July 2018 |
| | (The time-point when approximately 1000 dabigatran treated patients with completed observation time are expected to be registered in the database and data extraction will be done for the analysis) |
| Registration in the EU PAS register | 13 July 2017 (registration no. EUPAS 17165) |
| Final report of study results: | 31 December 2018 |
| | (Considering that the observation time for 1000 dabigatran treated patients is completed by 31 July 2018.) |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7. RATIONALE AND BACKGROUND

Stroke is the third most common cause of death in industrialised countries after myocardial infarcts and tumour diseases. [P90-55974] Stroke is also the most common cause of permanent disability. About 85% of all strokes are ischaemic, the remaining part haemorrhagic. One year after a total anterior circulation infarct, 60% of the patients have died and 35% have so severe neurological deficits that independent activities of daily living are restricted. With milder strokes, about 40% die or remain dependent. [R96-0250] Since the incidence of stroke is strongly age-related, the number of stroke victims is expected to increase substantially over the next decades when the proportion of the population over the age of 70 is estimated to grow from about 13% to 20%. Even within the next decade, the number of stroke victims is expected to increase by about 15%. [R17-1269]

The burden of stroke is heavy for the victims and for society. The yearly direct and indirect costs for stroke in Europe can be estimated to about 25 billion Euros. Since the stroke incidence is expected to be about 750.000 in ten years, these costs might increase by about 10-15% if we do not succeed to prevent more strokes and improve the effect of acute stroke intervention.

### Atrial fibrillation (AF) and stroke

Atrial fibrillation (AF) is the most common arrhythmia and the prevalence of AF is about 0.4 to 1% in the general population, rising to 8% in those subjects over 80 years. [R03-1233, R12-2675, P10-00760] The number of patients with AF is likely to increase 2.5-fold during the next 50 years. [R03-1233] Patients with AF have a 5 fold increased risk of ischemic stroke compared to persons without AF.[R96-0252] AF related strokes are more severe, are more likely to cause disability or to recur, and carry a higher mortality risk than strokes in patients without AF.[R09-4892, R10-0658, R10-0340] Clinical practice guidelines developed by the American College of Cardiology, American Heart Association, European Society of Cardiology, and American College of Chest Physicians recommend that all patients with AF and a CHADS₂ or CHA₂DS₂-VASc score ≥2 should receive long-term oral anticoagulation.[P10-10141, P11-03902, P12-01676] In the American College of Chest Physicians and European Society of Cardiology guidelines, oral anticoagulation also is recommended in patients with a CHADS<sub>2</sub> or CHA<sub>2</sub>DS<sub>2</sub>-VASc score of 1.[ P10-10141] Vitamin K antagonists (e.g. warfarin) were the only oral anticoagulants available until 2010 and updated guidelines include the newer oral anticoagulants as alternatives to vitamin K antagonists for stroke prevention. [P11-03902, P12-01676, P11-03903, P17-04650]

#### Anticoagulation treatment in patients with AF for stroke preventions

Long-term anticoagulation treatment reduces the incidence of ischemic stroke in patients with AF. In a meta-analysis, adjusted-dose warfarin reduced the risk of stroke by 64% compared to placebo and by approximately 40% compared to antiplatelet therapy.[P07-07953] Warfarin treatment is underused, particularly in elderly population and maintaining appropriate anticoagulation levels with warfarin is often difficult because of variable dose responses, multiple drug-drug and drug-food interactions, a slow onset and offset of action. Warfarin-treated patients require routine coagulation monitoring, dose adjustments, and dietary precautions to ensure a balance between therapeutic anticoagulation and bleeding risk.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Dabigatran, the first new Oral Anticoagulants

Dabigatran etexilate (Pradaxa) is the first non-Vitamin K Antagonist oral anticoagulant (NOAC) for stroke prevention in non-valvular atrial fibrillation (NVAF) patients. Dabigatran, a direct thrombin inhibitor, was evaluated in the phase III Randomized Evaluation of Longterm Anticoagulation Therapy (RE-LY) study. [P09-11669] Compared with warfarin, dabigatran 150 mg twice daily exhibited lower rates of stroke and systemic embolism, but similar rates of major haemorrhage; whereas treatment with dabigatran 110 mg twice daily showed similar rates of stroke and systemic embolism, but lower rates of major haemorrhage. Dabigatran has been approved more than 100 countries world-wide including Europe and US to reduce the risk of stroke and systemic embolism in patients with NVAF.

The European approved current version of Pradaxa® Summary of Product Characteristics (SmPC) can be found on the EMA Webpage:

• http://ec.europa.eu/health/documents/community-register/html/h442.htm.

The US approved version of the SmPC can be found on the FDA webpage:

 https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=overview.pr ocess&ApplNo=022512

Data from clinical studies such as RE-LY and RELY-ABLE [P09-11669, P13-08115] where the safety of dabigatran in stroke prevention has been demonstrated for up to 5 years were confirmed by studies in real world clinical practices in different patient populations. [P14-15648, P15-10687] However, it remains important to continue to address further real world clinical questions, which were so far not assessed in studies.

In RE-LY, severe, disabling stroke within the previous 6 months, or any stroke within the previous 14 days was excluded and therefore, data on the initiation of dabigatran treatment post-ischemic stroke for secondary stroke prevention in NVAF patients is sparse.

The initiation of warfarin for the secondary prevention of ischemic stroke in NVAF has been established over the years of its use and is based on the severity of the index event. It ranges between 2-3 days for TIA to 3-4 weeks for large ischemic insults. For dabigatran these initiation ranges after the index event have not yet been established. Therefore, the aim of this study is to explore the current real world use of dabigatran for stroke prevention in NVAF patients in the post-stroke setting. Therefore data on the timing of dabigatran treatment initiation will be described by analysing data on NVAF patients after hospitalization for acute ischemic stroke in this study.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8. RESEARCH QUESTION AND OBJECTIVES

### Primary objective:

• To evaluate the timing of dabigatran treatment initiation in patients with non-valvular atrial fibrillation (NVAF) after hospitalization for first ever ischaemic stroke (the index event), in order to prevent secondary stroke.

### Secondary objectives:

- To describe baseline characteristics for patients treated with dabigatran according to time of dabigatran initiation.
- To describe self-reported factors important for the physician's decision as to the time of dabigatran initiation in the post-ischemic stroke setting.
- To describe self-reported factors important for physician's decision as to which dabigatran dose was used in the post-ischemic stroke setting.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is an observational, multinational, multicentre, study in patients with NVAF presenting to a hospital with a first acute ischemic stroke. The study is based on existing data recorded in the SITS International Registry by physicians in European countries, such as Italy, United Kingdom, Czech Republic, Sweden, Germany, Poland, Spain, Finland, Portugal, Slovakia, Denmark, Estonia, Norway Belgium, Hungary, Slovenia, Croatia, Austria, Lithuania, France, Greece, Netherlands, Ireland, Ukraine and Iceland. All patients with NVAF will be included that present with the first ever ischemic stroke. For these patients baseline and demographics variables are available such as medical history including comorbidities and concomitant medications. Characteristics will further be used to estimate common stroke (CHADS<sub>2</sub>, CHA<sub>2</sub>DS<sub>2</sub>-VAS<sub>c</sub>) and bleeding (HAS-BLED) risk scores. Details on NVAF and secondary stroke prevention: time since first diagnosis, prior anticoagulation treatment, dose, and stroke severity of index event measured by National Institute of Health Stroke Scale (NIHSS) score, are recorded in the registry.

For patients that receive dabigatran within 3 months of the index event, details on post-stroke treatment (time from hospital admission – start and dose of dabigatran treatment for stroke prevention in NVAF, concomitant medication) will be analysed. Variables for physician's decision when to initiate oral anticoagulation with dabigatran post-ischemic stroke and the dose selected will be analysed.

In addition any start/stop of dabigatran treatment and doses prescribed will also be assessed at discharge and at 3 months after the index event.

### 9.2 SETTING

Patients with NVAF presenting with their first ever acute ischemic stroke who are registered in the SITS International Registry from 1 July 2014 until approximately 31 July 2018 will be included in the study.

#### **Inclusion criteria**

- Patients with non-valvular Atrial Fibrillation (NVAF)
- Patients presenting with their first acute ischemic stroke
- $\geq$  18 years of age

### **Exclusion criteria**

• Documentation that the patient was enrolled or is planned to be enrolled in an investigational clinical trial at the time of the onset of the index event and for the duration of the data collection

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9.3 VARIABLES

### 9.3.1 Exposures

Patient disposition will be provided according to post-stroke treatment (i.e. dabigatran, VKA, factor Xa inhibitors and no OAC therapy). Index event is defined as the acute ischemic stroke that led to hospital admission for eligible patients (baseline visit).

Dabigatran treated patients will be further stratified by newly diagnosed NVAF or prevalent NVAF, prior treatment with anticoagulation including type of anticoagulation therapy (dabigatran, VKA, Factor Xa Inhibitors, no anticoagulation) stroke severity measured by NIHSS score, dose of dabigatran, and timing of dabigatran treatment initiation. We will describe the timing of dabigatran treatment initiation for secondary prevention of stroke within 3 months after index event in the post-stroke setting. Timing of dabigatran treatment initiation will be summarized as a continuous variable as well as a categorical variable (see <a href="section 9.3.2.1">section 9.3.2.1</a>). For patients with dabigatran treatment initiated 28 days or more after index event, further analysis maybe carried out to determine their characteristics. These

#### 9.3.2 Outcomes

### 9.3.2.1 Primary outcomes

• The time lapsed from the index event to the initiation of the dabigatran treatment. This will be further categorized in specified time periods.

analyses will be detailed in a separate statistical analysis plan (see Appendix 4).

The following time periods will be considered, but could be revised (e.g. merging categories) depending on sample size 0-24h, >24-72h, >3-7d >7-14d, >14-28d, >28d-3m.

### 9.3.2.2 Secondary outcomes

- Description of baseline characteristics for patients treated with dabigatran according to time of dabigatran initiation.
- Description of self-reported factors important for physician's decision when to initiate dabigatran in the post-ischemic stroke setting for prevention of stroke and safety in NVAF.
- Description of self-reported factors important for physician's decision which dabigatran dose is used in the post-ischemic stroke setting for secondary prevention of stroke and safety in NVAF.

c03412460-01

#### **Definitions**

Ischemic stroke is defined as an event characterised by sudden onset of acute focal neurological deficit (e.g. resulting in an impairment of speech, motor function, cognition, gazes, vision, and/or neglect) presumed to be caused by cerebral ischemia/infarction after exclusion of haemorrhage by imaging scans.

The index event is the date of first ever ischemic stroke.

The 3 month follow-up data point for patients is 90 (+/- 10) days after the index event.

Major intracranial haemorrhage is defined as symptomatic intracranial bleeding at any time after start of dabigatran treatment and within 3 months from index event.

The evaluation of intracranial haemorrhage will be done using the available CT/MRI scan after start of dabigatran treatment and within 3 months from index event.

Major extracranial haemorrhage is derived from safety documentation in the SITS registry.

Death is defined as all cause death.

#### 9.3.3 Covariates

Patient characteristics such as age, stroke severity,(according to NIHSS) comorbidities, CHADS<sub>2</sub>, CHA<sub>2</sub>DS<sub>2</sub>-VAS<sub>c</sub>) and bleeding (HAS-BLED) risk scores (see <u>appendices 1-3</u>), prior oral anticoagulation treatment (dabigatran, Factor Xa Inhibitors, VKA, no OAC therapy), are regarded as potential covariates.

Patient characteristics will be assessed at index stroke date.

### 9.4 DATA SOURCES

### SITS – International Stroke Treatment Registry (ISTR)

Data from the SITS-International AF registry will be extracted for the purpose of analysis. The SITS-International registry is an ongoing, prospective, internet-based, academic-driven, multinational, stroke register. All centres registering patients in the SITS registry are required to accept the basic rules of participating in registry: consecutive registration of all patients with stroke symptoms receiving alteplase (if the centre registers only patients treated with intravenous thrombolysis), irrespective of whether treatment was on- or off-label. If the centre registers all stroke patients in the registry, consecutive registration of all patients with

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

stroke symptoms is obligatory. Death is collected separately in the SITS registry; however it is linked to the other outcomes at the 3 month time point from the index event. Register data has some inherent limitations. One of the most important limitations is we do not have any regular monitoring for source data verification, although monitoring was done during the period when the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) was done [P07-00880]. In 2011-12, Karolinska Trial Alliance performed an independent monitoring of some selected Swedish centres and verified that data entered in the registry from these centres are accurate. Moreover, it is important to note that all results published based on SITS data with regard to baseline and demographic characteristics and outcome are comparable to other published data from randomised trials, registry data and centre data. SITS registry has a logical automatic validation system, which prevents the entry of erroneous or impossible data in the registry, to some extent. Regular checking of online report and prompt action by contacting centre is also a part of the work for SITS International Coordination members. Moreover, data are downloaded and cleaned regularly for scientific publications.

The SITS registry has implemented extended data entry for AF and oral anticoagulation since June 2014.

### Specification of data collection from the index stroke event

At baseline: Demographic data, NIHSS and pre-stroke mRS, blood pressure, laboratory values (plasma glucose, cholesterol, coagulation status, liver function, kidney function,) medical history including comorbidities and concomitant medication, results of imaging scans, CHADS<sub>2</sub>, CHA<sub>2</sub>DS<sub>2</sub>-VASc and bleeding risk by HAS-BLED scores.

At 24 hours: NIHSS score, blood pressure, laboratory and imaging scans if performed. During hospital stay: details of concomitant medications, additional imaging scans prior to start of dabigatran treatment, any start/stop/change dabigatran treatment any results of the imaging scans

At 7 day or discharge if occurred earlier than 7 days: Date/time discharge, NIHSS scores, blood pressure, type of stroke and AF, medications

SITS is an academic-driven, non-profit, international collaboration. It is an initiative by the medical profession aimed at driving excellence in acute and secondary stroke treatment, and to develop new knowledge and leading research.

### 9.5 STUDY SIZE

Approximately 1000 NVAF patients who are treated with dabigatran etexilate within 3 months of index event constitute the main analysis population.

In order to address the further objective on characterisation of NVAF, the analysis population will be broadened to include all European patients with NVAF aged ≥18 presenting with their first acute ischemic stroke, regardless of subsequent oral anticoagulation use within the time period until approximately 1000 dabigatran patients are registered in SITS-AF.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Data will be extracted from the SITS-AF registry from the European dataset for retrospective analysis. The number of patients included in the study is not driven by a formal sample size calculation but rather by available patient numbers, only descriptive or exploratory analyses will be performed for this study.

### 9.6 DATA MANAGEMENT

Data in the SITS registry are entered on-line through the SITS website.

Each investigator/study nurse has a personal access code which must be kept secret and used only by the owner. All data entry from a centre can be made by each member of the local team, but once the data entry is confirmed (i.e., cannot be changed), the person who made the confirmation will be identified on the data entry form.

For the purpose of analysis, a download will be made in Excel/ CSV format which will then be transferred in the appropriate advance data analysis software such as STATISTICA/ SAS.

#### 9.7 DATA ANALYSIS

Descriptive statistics (absolute and relative frequencies, means, standard deviations, medians, inter quartile ranges, minimum and maximum values, 95% confidence intervals and proportions, as appropriate) for baseline and demographic characteristics for all included patients will be provided.

For the baseline characteristics we will calculate percentage proportions by dividing the number of events by the total number of patients, excluding missing or unknown cases as we generally did for all previous SITS-MOST and/or SITS-ISTR publications [P07-00880, P08-11746].

In the separate statistical analysis plan further sensitivity analyses may be added (see Appendix 4).

### 9.7.1 Main analysis

The main analysis will focus on NVAF patients presenting with first ischemic acute stroke and treated with dabigatran within 3 months of index event:

For patients initiated on dabigatran within 3 months of index event, the time to dabigatran treatment initiation will be summarized as a continuous variable as well as categorical; the following time periods will be considered, but could be revised (e.g. merging categories) depending on sample size 0-24h, >24-72h, >3-7d >7-14d, >14-28d, >28d-3m.

There will be a descriptive analysis of self-reported factors important for physicians decision when to initiate dabigatran and which dose in the post-ischemic stroke setting for prevention of stroke and safety in NVAF. This analysis will be done overall as well as by timing and by dose of dabigatran, respectively.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In addition, baseline and demographic characteristics will be presented stratified by timing and dose of dabigatran as well as by newly diagnosed NVAF or prevalent NVAF, prior treatment with anticoagulation including type of anticoagulation therapy, stroke severity measured by NIHSS score, if the sample size allows. Timing and dose of dabigatran treatment initiation will additionally the summarized for relevant baseline subgroups, e.g. based on stroke severity, if the sample size allows.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9.7.3 Interim analysis

Not applicable.

### 9.8 QUALITY CONTROL

The automatic quality control of data is included in the SITS-Registry. This includes immediate feedback if data are missing, out of range data, illogical or potentially erroneous data. In addition to automatic quality control, regular online data monitoring is performed by SITS International Coordinating Office (ICO) members. All changes in the registry are automatically logged in the database

In addition to online data monitoring, raw data are downloaded every 6 months to check for inconsistency, completeness. Normally investigators are informed by newsletter regarding the completeness of data entry for overall registry and asked to complete the missing data. In case of major inconsistency or high rate of missing data investigators are contacted personally by e-mail.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

### Non-interventional study based on existing data

The quality of a study based on existing data relies on accuracy of recorded data. Important data may not be available. In the absence of randomisation and blinding, it can be difficult to control for bias and confounders.

#### **Selection bias**

There is a risk of selection bias at the patient level. Sites might preferentially include "interesting" cases to the SITS study. To minimize selection bias at the patient level, centres were reminded by e-mail every 3 months that all consecutive patients from each site who meet entry criteria must be included in the SITS-Registry.

#### Lost to follow up

As with all observational studies a loss to follow up can occur. In this study this will affect the patients with a pre-planned follow up (patients initiating dabigatran within the 3 months after the index event). However, considering the short time period of the follow up and the lost to follow up at 3 months in the general SITS Registry being 20%, a similar percentage of lost to follow up is expected in this study as well.

### **Channeling bias**

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Channeling bias can occur due to preferential prescribing in relation to different risks for the events of interest: e.g., if dabigatran would be more often prescribed to higher risk patients compared to other treatments,

In order to assess potential channeling bias patients not receiving dabigatran within 3 months of the index event will be assessed. For example, patients initiating VKAs, other NOACs or no oral anticoagulation therapy will be assessed according to important patient baseline characteristics (e.g. age, sex, comorbidities, stroke and bleeding risk scores, concomitant medications).

### Confounding

As in any observational study, confounding may affect the estimation of association between variables and clinical outcome events of interest and statistical techniques such as adjustment for covariates, stratified analyses, matching, etc. can be used to correct for these. But as only major confounders for selected research questions can be captured, unmeasured confounding may remain.

#### **Exploratory analyses**

No formal power calculation has been done for this descriptive study and up to 1,000 patients with an index stroke are planned to be included. Follow-up is limited to three months after index stroke. Subgroup analyses, in particular those restricted to dabigatran patients, are only exploratory in nature. Exploratory analyses are usually not the definitive answer to the question at hand, but can be useful to define hypotheses to be tested in subsequent confirmatory studies.

### 9.10 OTHER ASPECTS

#### 9.10.1 Ethical approval and informed consent

The Institutional Review Board (IRB) or Independent Ethics Committee (IEC) of the Regional Ethical Review Board in Stockholm, Sweden (see website www.epn.se/en) has given approval for the SITS-Monitoring Study II (SITS-MOST II) protocol. SITS-MOST II is an 'over-arching' protocol that describes all research and analyses that SITS international is performing with the collected data in the SITS Registry, including this study 1160.235 (a part of the SITS-AF protocol in the SITS Registry).

The appendices in the SITS-MOST II protocol also include a patient information and informed consent form, describing the purpose of the SITS Registry and the reason why the patient is asked to collect their medical data in the SITS registry (see also Section 10).

The SITS-MOST II protocol and the EC approval document will be archived in the electronic Trial Master File (TMF), see <u>Appendix 4</u>.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9.11 SUBJECTS

Patients with non-valvular Atrial Fibrillation (NVAF) presenting with their first acute ischemic stroke and 18 years or older are study subject (see Section 9.2).

### 9.12 **BIAS**

To assess potential channeling bias baseline characteristics of all patients fulfilling the in/exclusion criteria and were included in SITS-AF registry in the defined time period will be described based on the treatment they receive for stroke prevention in NVAF within 3 months of the index event.

Differences in the patients that are initiated with dabigatran versus patients initiating with VKA, Factor Xa Inhibitors or no oral anticoagulation therapy will be described and set in context to the observed results in the dabigatran treated patient set (see also Section 9.9).

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10. PROTECTION OF HUMAN SUBJECTS

All data entered into the SITS International AF registry are encrypted in order to maintain patient data privacy. The individual patient and its research data is identified by a unique registry identification number. Access to data is strictly controlled by permitting each user a unique username and password. Additionally, each user has restrictions in viewing data sets, depending on their activity role in the database. Each data entry is centrally monitored by internal quality checks, such as automatic range checks and a full audit trail is maintained.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

According to the European Medicines Agency (EMA) Guideline on Good Pharmacovigilance Practices (GVP), Adverse Event (AE) reporting is not required for Non-Interventional Study (NIS) which is based on secondary data use.

As an observational study, based on existing data, all patient data is de-identified and will be analysed in aggregate. Individual patient safety related information will not be captured during this study. Thus, individual safety reporting is not applicable. Safety reporting will be done cumulatively in aggregate in the study report.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

After finalisation of the final report, manuscripts based on the results of the study are planned to be submitted to peer-reviewed medical journals. The steering committee will appoint a writing committee who will publish the manuscripts in the name of all investigators. A list of all investigators will be included in the original manuscript.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 13. REFERENCES

### 13.1 PUBLISHED REFERENCES

- P90-55974 WHO Task Force. Stroke-1989. Recommendations on stroke prevention, diagnosis and therapy. Report of the WHO Task Force on Stroke and other Cerebrovascular Disorders. Stroke 20 (10): 1407-1431 (1989)
- P06-10925 Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation.

  JAMA 285 (22), 2864 2870 (2001)
- P07-00880 Wahlgren N, Ahmed N, Davalos A, et al. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet 369 (9558): 275-282 (2007)
- P07-07953 Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have non-valvular atrial fibrillation. Ann Intern Med, 146 (12), 857–867 (2007)
- P08-11746 Wahlgren N, Ahmed N, Davalos A, et al. Thrombolysis with alteplase 3-4.5 h after acute ischaemic stroke (SITS-ISTR): an observational study. Lancet 372 (9646):1303-1309 (2008)
- P09-11669 Connolly SJ, Ezekowitz MD, Yusuf S, et al. (RE-LY study). Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med, 361 (12), 1139–1151 (2009)
- P10-00760 Fuster V, Ryden LE, Cannom DS, et al. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation 114: e257-354 (2006)
- P10-10141 Camm AJ, Kirchhof P, Lip GYH, et al. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J, 31 (19), 2369–2429 (2010)
- P11-03902 Wann LS, Curtis AB, Ellenbogen KA, et al. 2011 ACCF/AHA/HRS focused updates incorporated into the ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation: a report of the American

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation 123 (10), e269–e367 (2011) P11-03903 Wann LS, Curtis AB, Ellenbogen KA, et al. 2011 ACCF/AHA/HRS focused update on the management of patients with atrial fibrillation (update on dabigatran): a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol 57 (11), 1330–1337 (2011) P12-01676 You JJ, Singer DE, Howard PA, et al. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest 141 (2) (Suppl), e531S–e575S (2012) P13-08115 Connolly SJ, Wallentin L, Ezekowitz MD, et al. The Long Term Multi-Center Observational Study of Dabigatran Treatment in Patients with Atrial Fibrillation: (RELY-ABLE) Study. Circulation 128 (3), 237-243 (2013) P14-15648 Graham DJ, Reichman ME, Wernecke M, Zhang R, Southworth MR, Levenson M, Sheu TC, Mott K, Goulding MR, Houstoun M, MaCurdy TE, Worrall C, Kelman JA. Cardiovascular, bleeding, and mortality risks in elderly Medicare patients treated with dabigatran or warfarin for non-valvular atrial fibrillation. Circulation 131 (2), 157–164 (2015) P15-10687 Villines TC, Schnee J, Fraeman K, Siu K, Reynolds MW, Collins J, Schwartzman E. A comparison of the safety and effectiveness of dabigatran and warfarin in non-valvular atrial fibrillation patients in a large healthcare system. Thromb Haemost. 114 (6), 1290-1298 (2015) P17-04650 Shahid F, Shantsila E, Lip GYH. What do the guidelines suggest for nonvitamin K antagonist oral anticoagulant use for stroke prevention in atrial fibrillation? Eur Heart J 18 (Suppl I), 118-124 (2016) R96-0250 Bamford J, Sandercock P, Dennis M, Burn J, Warlow C. Classification and natural history of clinically identifiable subtypes of cerebral infarction. Lancet 337 (8756, 1521-1526 (1991) Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk R96-0252 factor for stroke: the Framingham Study. Stroke 22 (8), 983-988 (1991) Go AS, Hylek EM, Phillips KA, et al. Prevalence of diagnosed atrial R03-1233 fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA 285 (18), 2370-2375 (2001) Lin HJ, Wolf PA, Kelly-Hayes M, et al. Stroke severity in atrial fibrillation. R09-4892 The Framingham Study. Stroke 27 (10), 1760–1764 (1996)

c03412460-01

| R10-0340 | Dulli DA, Stanko H, Levine RL. Atrial fibrillation is associated with severe acute ischemic stroke. Neuroepidemiology 22 (2), 118–123 (2003) |
|---|---|
| R10-0658 | Jorgensen HS, Nakayama H, Reith J, et al. Acute stroke with atrial fibrillation. The Copenhagen Stroke Study. Stroke, 27 (10), 1765–1769 (1996) |
| R10-5332 | Lip GYH, Nieuwlaat R, Pisters R, Lane DA, Crijns HJGM. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the Euro Heart Survey on Atrial Fibrillation. Chest 137 (2), 263 - 272 (2010) |
| R10-6394 | Pisters R, Lane DA, Nieuwlaat R, Vos CB de, Crijns HJGM, Lip GYH A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest 138 (5), 1093 - 1100 (2010) |
| R12-2675 | Furberg CD, Psaty BM, Manolio TA, et al. Prevalence of atrial fibrillation in elderly subjects (the Cardiovascular Health Study). Am J Cardiol 74 (3), 236-241 (1994) |
| R17-1269 | Wahlgren NG. Introduction. In: Wahlgren NG, editor. Update on Stroke Therapy 2000-2001, Stockholm: Karolinska Stroke Update, 17-19 (2001) |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 14. APPENDICES

### APPENDIX 1: CHADS<sub>2</sub> STROKE RISK SCORE

| CHADS <sub>2</sub> components | Points |
|---------------------------------------------|--------|
| Congestive heart failure | 1 |
| Hypertension | 1 |
| Age 75 years or older | 1 |
| Diabetes mellitus | 1 |
| Prior cerebral ischemia (i.e., stroke, TIA) | 2 |
| Maximum score | 6 |

CHADS<sub>2</sub> score is based on a point system in which 2 points are assigned for a history of stroke or transient ischemic attack and 1 point each is assigned for age 75 years or older, hypertension, diabetes, or clinical heart failure or impaired left ventricular systolic function (generally interpreted as an ejection fraction  $\leq 40\%$ ). A CHADS<sub>2</sub> score of 0 identifies patients at low stroke risk, a score of 1 to 2 identifies patients at moderate stroke risk, and a score greater than 2 identifies patients at high stroke risk [P06-10925].

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### APPENDIX 2: CHA2DS2-VASC STROKE RISK SCORE

| CHA <sub>2</sub> DS | <sub>2</sub> VAS <sub>c</sub> score | |
|---|---|---|
| Risk factors for stroke and thro | mbo-embolism in non | -valvular AF |
| Major risk factors | Clinically releva | · · |
| Previous stroke, TIA, or systemic embolism Age ≥ 75 years | Heart failure or moderate to severe LV systolic dysfunction (e.g. LV EF <40 %) Hypertension - Diabete mellitus Female sex - Age 65-74 years Vascular disease | |
| Risk factor-based approach expression with the acrony (Note: maximum score is 9 since | ym CHA <sub>2</sub> DS <sub>2</sub> -VAS <sub>c</sub> | |
| Risk factor | age may contribute 0, | Score |
| Congestive heart failure/LV dysfund | ction | 1 |
| Hypertension | | 1 |
| Age ≥75 | | 2 |
| Diabetes mellitus | | 1 |
| Stroke/TIA/systemic embolism | | 2 |
| Vascular disease* | | 1 |
| Age 65-74 | | 1 |
| - | | |

Sex category (i.e. female sex)

Maximum score

The CHA<sub>2</sub>DS<sub>2</sub>-VASc risk score is based on a point system in which 2 points are assigned for a history of stroke or TIA, or age  $\geq$ 75; and 1 point each is assigned for age 65–74 years, a hypertension, diabetes, cardiac failure, vascular disease and female sex. On the basis of the risk strata defined in previous guidelines, a CHA<sub>2</sub>DS<sub>2</sub>-VASc score of 0 corresponds to "low risk", a score of 1 corresponds to "intermediate risk", and a score of 2 or more corresponds to "high risk" [R10-5332].

1

9

<sup>\*</sup> Myocardial infarction, complex aortic plaque and PAD

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### APPENDIX 3: HAS-BLED BLEEDING RISK SCORE

| Clinical | l characteristics comprising the HAS-I | BLED bleeding risk |
|---|---|---|
| Letter | Clinical characteristic | Points awarded |
| Н | Hypertension | 1 |
| A | Abnormal renal and liver function (1 point each) | 1 or 2 |
| S | Stroke | 1 |
| В | Bleeding | 1 |
| L | Labile INRs | 1 |
| Е | Elderly (e.g. age >65 years) | 1 |
| D | Drugs or alcohol (1 point each) | 1 or 2 |
| Maxi | mum score | 9 |

Hypertension is defined as history of hypertension and current uncontrolled systolic blood pressure >160 mmHg. 'Abnormal kidney function' is defined as the presence of chronic dialysis or renal transplantation or serum creatinine  $\geq$ 200  $\mu$ mol/L. 'Abnormal liver function' is defined as chronic hepatic disease (e.g. cirrhosis) or biochemical evidence of significant hepatic derangement (e.g. bilirubin >2 x upper limit of normal, in association with aspartate aminotransferase/alanine aminotransferase/alkaline phosphatase >3 x upper limit normal). 'Bleeding' refers to previous bleeding history and/or predisposition to bleeding, e.g. bleeding diathesis, anaemia, etc. 'Labile INRs' refers to unstable/high INRs or poor time in therapeutic range (e.g. <60%). Drugs/alcohol use refers to concomitant use of drugs, such as antiplatelet agents, non-steroidal anti-inflammatory drugs, or alcohol abuse, etc. If a patient is not on VKA the value for 'labile INRs' will be set to 0. Further details will be given in the separate statistical analysis plan (see <u>Appendix 4</u>).

A HAS-BLED score of  $\geq 3$  indicates 'high risk' for AF patients to develop a bleed and some caution and regular review of the patient is needed following the initiation of antithrombotic therapy, whether with VKA or aspirin [R10-6394].

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **APPENDIX 4: LIST OF STAND-ALONE DOCUMENTS**

The final version of the following stand-alone documents will be archived in the Trial Master File (TMF)

- Statistical analysis plan (and revisions, if applicable)
- SITS-MOST II protocol (and amendments, if applicable)
- Ethics Committee approval(s) for the SITS-MOST II protocol (and amendments, if applicable)

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### APPENDIX 5: ENCEPP CHECKLIST FOR STUDY PROTOCOLS





Doc.Ref. EMA/540136/2009

European Network of Centres for Pharmacoepidemiology and Pharmacovigilance

#### **ENCePP Checklist for Study Protocols (Revision 3)**

Adopted by the ENCePP Steering Group on 01/07/2016

The <u>European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP)</u> welcomes innovative designs and new methods of research. This Checklist has been developed by ENCePP to stimulate consideration of important principles when designing and writing a pharmacoepidemiological or pharmacovigilance study protocol. The Checklist is intended to promote the quality of such studies, not their uniformity. The user is also referred to the <u>ENCePP Guide on Methodological Standards in Pharmacoepidemiology</u>, which reviews and gives direct electronic access to guidance for research in pharmacoepidemiology and pharmacovigilance.

For each question of the Checklist, the investigator should indicate whether or not it has been addressed in the study protocol. If the answer is "Yes", the section number of the protocol where this issue has been discussed should be specified. It is possible that some questions do not apply to a particular study (for example, in the case of an innovative study design). In this case, the answer 'N/A' (Not Applicable) can be checked and the "Comments" field included for each section should be used to explain why. The "Comments" field can also be used to elaborate on a "No" answer.

This Checklist should be included as an Annex by marketing authorisation holders when submitting the protocol of a non-interventional post-authorisation safety study (PASS) to a regulatory authority (see the <u>Guidance on the format and content of the protocol of non-interventional post-authorisation safety studies</u>). The Checklist is a supporting document and does not replace the format of the protocol for PASS as recommended in the Guidance and Module VIII of the Good pharmacovigilance practices (GVP).

Study title: Pradaxa Initiation Post-Stroke Study: SITS-Pradaxa 1. An analysis from the SITS-AF Registry on treatment initiation of dabigatran etexilate in non-valvular atrial fibrillation patients hospitalized with acute ischemic stroke

#### Study reference number: 1160-0235

| Sec | tion 1: Milestones | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 1.1 | Does the protocol specify timelines for | | | | |
| | 1.1.1 Start of data collection <sup>1</sup> | | | | 6 |
| | 1.1.2 End of data collection <sup>2</sup> | | | | 6 |
| | 1.1.3 Study progress report(s) | | | $\boxtimes$ | * |
| | 1.1.4 Interim progress report(s) | | | $\boxtimes$ | 9.7.3 |
| | 1.1.5 Registration in the EU PAS register | | | | 6 |
| | 1.1.6 Final report of study results. | | | | 6 |

Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts.

<sup>2</sup> Date from which the analytical dataset is completely available.

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | ments: | | | | |
|---|---|---|---|---|---|
| Sec | tion 2: Research question | Yes | No | N/A | Section<br>Number |
| 2.1 | Does the formulation of the research question and objectives clearly explain: | | | | 8 |
| | 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) | ⊠ | | | 7 |
| | 2.1.2 The objective(s) of the study? | $\boxtimes$ | | | 8 |
| | 2.1.3 The target population? (i.e. population or subgroup<br>to whom the study results are intended to be generalised) | ⊠ | | | 9.2 |
| | 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | $\boxtimes$ | See comment |
| | 2.1.5 If applicable, that there is no a priori hypothesis? | | | | 9.9 |
| Com | ments: | | | | |
| 2.1.4 | . Descriptive statistical analysis only | | | | |
| Sect | tion 3: Study design | Yes | No | N/A | Section<br>Number |
| 3.1 | Is the study design described? (e.g. cohort, case-<br>control, cross-sectional, new or alternative design) | | | | 9.1 |
| 3.2 | Does the protocol specify whether the study is<br>based on primary, secondary or combined data<br>collection? | $\boxtimes$ | | | 9.9,<br>11 |
| 3.3 | Does the protocol specify measures of occurrence? (e.g. incidence rate, absolute risk) | | | | 9.3.2.3,<br>9.7.2 |
| 3.4 | Does the protocol specify measure(s) of association? (e.g. relative risk, odds ratio, excess risk, incidence rate ratio, hazard ratio, number needed to harm (NNH) per year) | | | × | |
| 3.5 | Does the protocol describe the approach for the collection and reporting of adverse events/adverse reactions? (e.g. adverse events that will not be collected in case of primary data collection) | × | | | 11 |
| Com | ments: | | · . | | |
| 3.5 I<br>done | ndividual safety reporting (AE collection) will not be done in<br>in aggregated fashion. | this obs | ervation | nal study | , but will be |
| Sect | ion 4: Source and study populations | Yes | No | N/A | Section<br>Number |
| 4.1 | Is the source population described? | Ø | | | 9.2,<br>9.4,<br>9.5 |
| 4.2 | Is the planned study population defined in terms of: | | | | |
| | 4.2.1 Study time period? | | | | 6 |
| | 4.2.2 Age and sex? | $\boxtimes$ | | | 9.2 |

**ENCePP Checklist for Study Protocols (Revision 3)** 

c03412460-01

| Sec | tion 4: Source and study populations | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| | 4.2.3 Country of origin? | | | | 9.1 |
| | 4.2.4 Disease/indication? | $\boxtimes$ | | | 9.2 |
| | 4.2.5 Duration of follow-up? | | | | 9.1 |
| 4.3 | Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | × | | | |
| Com | ments: | | | | |
| Sec | tion 5: Exposure definition and measurement | Yes | No | N/A | Section<br>Number |
| 5.1 | Does the protocol describe how the study exposure is defined and measured? (e.g. operational details for defining and categorising exposure, measurement of dose and duration of drug exposure) | ⊠ | | | 9.3.1,<br>9.7.2 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation sub-study) | | | | 9.4,<br>9.8<br>+see comment |
| 5.3 | Is exposure classified according to time windows? (e.g. current user, former user, non-use) | ⊠ | | | 9.7.2 |
| 5.4 | Is exposure classified based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | ⊠ | |
| 5 | ments: i.2: sections 9.4 (Data sources) and 9.8 (Quality control) incorposure. | directly a | ddresse | s the m | easurement of |
| Sect | ion 6: Outcome definition and measurement | Yes | No | N/A | Section<br>Number |
| 6.1 | Does the protocol specify the primary and<br>secondary (if applicable) outcome(s) to be<br>investigated? | ⊠ | | | 8, |
| 6.2 | Does the protocol describe how the outcomes are defined and measured? | | | | 8, 9.3.2 |
| 6.3 | Does the protocol address the validity of outcome<br>measurement? (e.g. precision, accuracy, sensitivity,<br>specificity, positive predictive value, prospective or<br>retrospective ascertainment, use of validation sub-study) | ⊠ | | | 9.4,<br>9.8<br>+see comment |
| 6.4 | Does the protocol describe specific endpoints relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease, disease management) | | ⊠ | | |
| Com | ments: | | | | |
| | sections 9.4 (Data Sources) and 9.8 (Quality Control) indire | ctly addr | esses th | ne outco | me |

c03412460-01

| Sec | tion 7: Bias | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 7.1 | Does the protocol describe how confounding will be addressed in the study? | Ø | | | 9.9 |
| | 7.1.1. Does the protocol address confounding by indication if applicable? | | | | See commen |
| 7.2 | Does the protocol address: | | - | | |
| | 7.2.1. Selection biases (e.g. healthy user bias) | $\boxtimes$ | | | 9.9 |
| | <ol> <li>7.2.2. Information biases (e.g. misclassification of<br/>exposure and endpoints, time-related bias)</li> </ol> | | $\boxtimes$ | | See commen |
| 7.3 | Does the protocol address the validity of the study covariates? | | | | 9.3.3 |
| Com | iments: | | | | |
| 5tud<br>7.2.: | 2: Selection bias, lost to follow up and channeling bias are de | escribed | | | |
| Sec | tion 8: Effect modification | Yes | No | N/A | Section<br>Number |
| 8.1 | Does the protocol address effect modifiers?<br>(e.g. collection of data on known effect modifiers, sub-group<br>analyses, anticipated direction of effect) | | | × | , and a |
| Com | ments: | | | | |
| This | descriptive study does not assess treatment effects. | | | | |
| Sec | tion 9: Data sources | Yes | No | N/A | Section<br>Number |
| 9.1 | Does the protocol describe the data source(s) used<br>in the study for the ascertainment of: | | | | |
| | 9.1.1 Exposure? (e.g. pharmacy dispensing, general<br>practice prescribing, claims data, self-report, face-to-face<br>interview) | $\boxtimes$ | | | 9.1, |
| | 9.1.2 Outcomes? (e.g. clinical records, laboratory markers<br>or values, claims data, self-report, patient interview<br>including scales and questionnaires, vital statistics) | $\boxtimes$ | | | 8,<br>9.4 |
| | 9.1.3 Covariates? | $\boxtimes$ | | | 9.3.3, |
| | | | 10000 | 100 | 9.9 |
| 9.2 | Does the protocol describe the information available from the data source(s) on: | | | | 9.9 |
| 9.2 | | × | | | 9.9<br>9.1,<br>9.4 |
| 9.2 | available from the data source(s) on: 9.2.1 Exposure? (e.g. date of dispensing, drug quantity, dose, number of days of supply prescription, daily dosage, | ⊠<br>⊠ | | | 9.1, |
| 9.2 | available from the data source(s) on: 9.2.1 Exposure? (e.g. date of dispensing, drug quantity, dose, number of days of supply prescription, daily dosage, prescriber) 9.2.2 Outcomes? (e.g. date of occurrence, multiple event, | | | | 9.1,<br>9.4<br>9.1,<br>9.3.2, |

c03412460-01

| Sect | tion 9: Data sources | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| | 9.3.1 Exposure? (e.g. WHO Drug Dictionary, Anatomical<br>Therapeutic Chemical (ATC) Classification System) | | × | | |
| | 9.3.2 Outcomes? (e.g. International Classification of<br>Diseases (ICD)-10, Medical Dictionary for Regulatory<br>Activities (MedDRA)) | | × | | |
| | 9.3.3 Covariates? | | $\boxtimes$ | | |
| 9.4 | Is a linkage method between data sources described? (e.g. based on a unique identifier or other) | | | | 10 |
| Com | ments: | | | 417 | |
| Sect | ion 10: Analysis plan | Yes | No | N/A | Section<br>Number |
| 10.1 | Is the choice of statistical techniques described? | | | | 9.6 |
| 10.2 | Are descriptive analyses included? | | | | 9.3.2.2,<br>9.5,<br>9.7 |
| 10.3 | Are stratified analyses included? | | | | 9.3.2,<br>9,7 |
| 10.4 | Does the plan describe methods for adjusting for confounding? | | | | |
| 10.5 | Does the plan describe methods for handling missing data? | | | | 9.7,<br>9.8 |
| 10.6 | Is sample size and/or statistical power estimated? | | | | 9.5<br>+see commer |
| Com | ments: | | | | |
| 10.6: | Statistical power is not assessed as no comparisons are pl | anned. | | | |
| Sect | ion 11: Data management and quality control | Yes | No | N/A | Section<br>Number |
| 11.1 | Does the protocol provide information on data<br>storage? (e.g. software and IT environment, database<br>maintenance and anti-fraud protection, archiving) | ⋈ | | | 9.6,<br>10 |
| 11.2 | Are methods of quality assurance described? | | | | 9.4,<br>9.8,<br>10 |
| 11.3 | Is there a system in place for independent review of study results? | ⊠ | | | 12 |
| Com | ments: | | | // | |
| Sect | ion 12: Limitations | Yes | No | N/A | Section<br>Number |
| 12.1 | Does the protocol discuss the impact on the study results of: | | | | |

c03412460-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Yes | No | N/A | Section<br>Number |
|---|---|---|---|
| $\boxtimes$ | | | 9.9 |
| | $\boxtimes$ | | |
| | | | 9.9 |
| | | × | 9.2,<br>9.3.1,<br>9.5, 9.9 |
| Yes | No | N/A | Section |
| | | | Number |
| | | | 9.10.1 |
| Ø | | | 9.10.1 |
| $\boxtimes$ | | | 10 |
| Yes | No | N/A | Section |
| | | | Number<br>5 |
| Yes | No | N/A | Section<br>Number |
| Yes | No | N/A | |
| 9550 | 100 | N/A | Number |
| | Yes Yes | Yes No Yes No Yes No | Yes No N/A Yes No N/A Yes No N/A |

ENCePP Checklist for Study Protocols (Revision 3)